CLINICAL TRIAL: NCT04214574
Title: Real-Time Ultrasound-Guided Neuraxial Puncture in Elderly Patients: A Randomized Controlled Trial Comparing Between Paramedian Transverse and Parasagittal Oblique
Brief Title: Real Time Ultrasound Guided Spinal Anesthesia in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Marwan Rizk, Principal Investigator, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2018-0589
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Realtime Ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of the study, blinding of the anesthesiologist was not possible
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real time ultrasound-guided Parasagittal oblique technique (RTU-PO) (Experimental): In the RTU-PO group, the probe will be placed in a parasagittal plane to identify the articular processes then the sacrum will be identified. The probe will be moved cephalad in the parasagittal axis until the identification of the target lumbar interspaces L2-L3, L3-L4 or L4-L5. Once the appropriate lumbar interspace is identified, the probe will be tilted 45 degree towards the midline into a parasagittal oblique view. This provides a view of the paramedian interlaminar space. The ligamentum flavum and the dura form the posterior complex that can be often visualized as a single hyperechoic structure beneath which lies the hypoechoic intrathecal space. The needle will be inserted in plane from the caudal end of the ultrasound transducer with its tip directed towards the interlaminar space under real-time in-plane US guidance.
  Interventions: Device: Parasagittal oblique technique (Ultrasound)
- Real time ultrasound-guided paramedian tranverse technique (RTU-T) (Experimental): In the RTU-T group, similar to the RTU-PO group, the transducer will be applied in the parasagittal plane, and after identification of the intervertebral level, the probe will be rotated 90 degrees into a transverse orientation and centered on the neuraxial midline in a way to align the beam with the interspinous and interlaminar space and thus to get a paramedian transverse interlaminar view. The needle will be inserted in plane from the lateral end of the ultrasound transducer with its tip directed towards the medial border of the articular process.
  Interventions: Device: Paramedian tranverse technique (Ultrasound)

INTERVENTIONS:
Device: Parasagittal oblique technique (Ultrasound) — the probe will be placed in a parasagittal plane to identify the articular processes then the sacrum will be identified. The probe will be moved cephalad in the parasagittal axis until the identification of the target lumbar interspaces L2-L3, L3-L4 or L4-L5. Once the appropriate lumbar interspace is identified, the probe will be tilted 45 degree towards the midline into a parasagittal oblique view. The needle will be inserted in plane from the caudal end of the ultrasound transducer with its tip directed towards the interlaminar space under real-time in-plane US guidance.
  Arms: Real time ultrasound-guided Parasagittal oblique technique (RTU-PO)
Device: Paramedian tranverse technique (Ultrasound) — the transducer will be applied in the parasagittal plane, and after identification of the intervertebral level, the probe will be rotated 90 degrees into a transverse orientation and centered on the neuraxial midline in a way to align the beam with the interspinous and interlaminar space and thus to get a paramedian transverse interlaminar view. The needle will be inserted in plane from the lateral end of the ultrasound transducer with its tip directed towards the medial border of the articular process.
  Arms: Real time ultrasound-guided paramedian tranverse technique (RTU-T)

SUMMARY:
In this prospective randomized observational study, investigators aim to compare the efficacy and procedural outcomes of real-time ultrasound guided parasagittal oblique (RTU-PO) and real-time ultrasound guided paramedian transverse (RTU-PT) approaches in elderly patients undergoing elective surgery under spinal anesthesia.

DETAILED DESCRIPTION:
Background: Since its first introduction in 1898 by Bier, Spinal anesthesia has been performed using the anatomical landmark guided approach. Despite being useful, the landmark technique doesn't take into account anatomical variations, spine abnormalities or age-related changes in the lumbar spine as seen in elderly, obese or pregnant patients and thus can lead to incorrect identification of a certain interspace. Neuraxial ultrasonography has been introduced as a technique to allow the operator to preview spinal anatomy, identify the midline, determine the interspace and guide the needle insertion site and trajectory. It was found to be a feasible and promising technique that can result in successful cerebrospinal fluid acquisition where other methods have failed. While pre-procedural Ultrasound has been used by many studies to identify the right epidural or subarachnoid spaces and have an idea about the angle of needle insertion, it remains a blind technique. Real-time ultrasound guided technique was found to improve the limitations of the pre-puncture ultrasound guided techniques by direct, real-time visualization of the needle trajectory. In spinal anesthesia, a midline approach has been the most common technique used for needle insertion. However, this approach is often technically difficult in the geriatric population because of poorly palpable surface landmarks, lumbar scoliosis, marked thoracic kyphosis, degenerative changes and inability to flex the lumbar spine in the sitting position. While the parasagittal oblique approach tends to provide a better sonographic window into the vertebral canal than the midline approach, it is still not evident whether it will lead to an easier paramedian needle insertion. In the literature, there are no studies directly comparing the paramedian transverse and parasagittal oblique approaches in the performance of real time ultrasound guided spinal anesthesia.

Specific Aim: The aim of this study is to find out the optimal approach to perform spinal anesthesia under real time ultrasound guidance in the elderly population. Thus, investigators will compare real time ultrasound-guided paramedian approach using parasagittal oblique view with real time ultrasound guided paramedian approach using the paramedian transverse median view. The aim is thus to adopt a real time ultrasound guided technique that will result in an easier access to the subarachnoid space in patients with difficult anatomy and results in better patient satisfaction and less discomfort.

Methodology and analysis: In a prospective randomized observational study, 84 patients scheduled for surgery amenable to spinal anesthesia, aged more than 65 years, with American Society of Anesthesiologists physical status 1 to 3 will be assigned to receive spinal anesthesia to one of two treatment groups: real time ultrasound-guided parasagittal oblique technique (group RTU-PO) or Real time ultrasound-guided paramedian transverse technique (group RTU-T). Ultrasonography of the lumbar spine and Real time spinal blockade will be performed by the experienced anesthesiologist. Patients in both groups will have an ultrasound scan of the lumbar spine to measure the depth of the dura, to specify and guide the needle insertion site and trajectory. The primary outcome is the rate of successful dural puncture on the first needle insertion attempt under real time ultrasound guidance. Normally distributed data will be summarized as mean ± SD and nonnormally distributed data will be summarized as median [interquartile range].

Significance: Investigators believe that real time US-guided technique is a superior modality of performance of spinal anesthesia. However, investigators would like to evaluate which approach will be better for the acquisition of cerebrospinal fluid in elderly patients. Investigators think that this study would have an impact on current practice in term of introducing real time ultrasound guided technique into everyday practice and determining the best approach to perform a successful neuraxial block in a patient with a suspected difficult back.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging above 65 years
* American Society of Anesthesiologists physical status 1 to 3
* Can give informed consent
* Scheduled for elective surgery

Exclusion Criteria:

* Inability to sit or to give consent
* Patients with severe cardiopulmonary diseases
* Previous back surgery or spinal congenital abnormalities
* Bleeding diathesis
* Anticoagulants or antiplatelets except aspirin
* Local anesthesia allergy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Incidence of successful Dural puncture on the first needle insertion attempt | At the begining of the procedure (during the needle insertion)
  Successful needle insertion on the first attempt (Yes/No)

SECONDARY OUTCOMES:
Incidence of success of spinal anesthesia | During the procedure
  Success of spinal anesthesia (Yes/No)
Time to identify posterior complex on ultrasound | During the procedure
  Time to identify posterior complex on ultrasound (measured in seconds)
Time to perform spinal anesthesia | During the procedure
  Time to perform spinal anesthesia (measured in seconds)
Procedural time | During the procedure
  Procedural time (measured in minutes)
Depth of the posterior complex | During the procedure
  Depth of the posterior complex (measured in cm)
Number of redirections | During the procedure
  Number of redirections
Number of needle passes | During the procedure
  Number of needle passes
Number of separate skin punctures | During the procedure
  Number of separate skin punctures
Number of spinal levels attempted | During the procedure
  Number of spinal levels attempted
Rate of satisfaction | After the procedure
  Patient satisfaction (scale from 1 to 3: very satisfied, satisfied, dissatisfied)
Rate of complications | During the procedure
  Complications (Yes/No)
Rate of complications, if present | During the procedure
  Complications if present (Vascular puncture, Paresthesia, Conversion to GA 30 minutes after block, and Others)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Rizk, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon